CLINICAL TRIAL: NCT01168297
Title: Type 2 Diabetes and Obesity in Mexican Pimas: Gene-Environment Interaction
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910161; 10-DK-N161
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Obesity; Type 2 Diabetes Mellitus; Genetics; Energy Expenditure; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Maycoba residents: Pima and non-Pima Mexicans from the village of Maycoba

SUMMARY:
In 1995 we conducted a cross-sectional study to identify the effects of traditional and western environments on prevalence of type 2 diabetes mellitus (T2DM) and obesity in Pima Indians in Mexico and the United States. The Mexican Pimas live in a remote mountainous region and at that time had experienced little change from their traditional lifestyle. Nothing was known about their T2DM prevalence. A similar number of non-Pima Mexicans live in the same village. In contrast to the Mexican Pimas, the U.S. Pimas live in more westernized society and have a high prevalence of diabetes. We found that although T2DM and obesity were more prevalent in Mexican Pimas than non-Pimas, both Mexican groups had a significantly lower prevalence of these disorders than U.S. Pimas. The lifestyle of the Mexican population studied included a dramatically higher level of physical activity and a diet higher in fiber and lower in calories derived from fat compared with the U.S. Pimas. Since the U.S. and Mexican Pimas share a similar gene pool we concluded that even in populations genetically prone to T2DM and obesity, their development is determined largely by environmental circumstances.

Since 1995 the environmental circumstances of the Mexican Pimas and non-Pimas have changed. The electrical supply to the region has increased, cars have become more prevalent and grocery stores have appeared. The impact of these changes on T2DM and obesity has not been examined. In light of these events, we propose to: 1) compare the current prevalence of T2DM and obesity in Mexican Pimas and non-Pima Mexicans to that present in 1995 with the same measures used previously, including height, weight, waist circumference, body composition by bioelectrical impedance, oral glucose tolerance and HbA1c; 2) compare current diet, physical activity and total energy expenditure in both Mexican Pimas and. non-Pima Mexicans using the same methods as the 1995 study to the previous results and 3) document the frequencies of T2DM and obesity-associated genetic variants in Mexican Pimas compared with U.S. Pimas and non-Pima Mexicans.

DETAILED DESCRIPTION:
In 1995 we conducted a cross-sectional study to identify the effects of traditional and western environments on prevalence of type 2 diabetes mellitus (T2DM) and obesity in Pima Indians in Mexico and the United States. The Mexican Pimas live in a remote mountainous region and at that time had experienced little change from their traditional lifestyle. Nothing was known about their T2DM prevalence. A similar number of non-Pima Mexicans live in the same village. In contrast to the Mexican Pimas, the U.S. Pimas live in more westernized society and have a high prevalence of diabetes. We found that although T2DM and obesity were more prevalent in Mexican Pimas than non-Pimas, both Mexican groups had a significantly lower prevalence of these disorders than U.S. Pimas. The lifestyle of the Mexican population studied included a dramatically higher level of physical activity and a diet higher in fiber and lower in calories derived from fat compared with the U.S. Pimas. Since the U.S. and Mexican Pimas share a similar gene pool we concluded that even in populations genetically prone to T2DM and obesity, their development is determined largely by environmental circumstances.

Since 1995 the environmental circumstances of the Mexican Pimas and non-Pimas have changed. The electrical supply to the region has increased, cars have become more prevalent and grocery stores have appeared. The impact of these changes on T2DM and obesity has not been examined. In light of these events, we propose to: 1) compare the current prevalence of T2DM and obesity in Mexican Pimas and non-Pima Mexicans to that present in 1995 with the same measures used previously, including height, weight, waist circumference, body composition by bioelectrical impedance, oral glucose tolerance and HbA1c; 2) compare current diet, physical activity and total energy expenditure in both Mexican Pimas and. non-Pima Mexicans using the same methods as the 1995 study to the previous results and 3) document the frequencies of T2DM and obesity-associated genetic variants in Mexican Pimas compared with U.S. Pimas and non-Pima Mexicans.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Selection of Subjects:

-The entire adult population of Maycoba, Sonora, Mexico, will be invited to participate in the main study. Individuals will be eligible to participate if they are at least 18 years old and residents of Maycoba and able to give informed consent. There will be no further exclusion or inclusion criteria. For the doubly-labeled water studies pregnant women will be excluded, since pregnancy has profound effects on energy expenditure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of Maycoba, Sonora, Mexico@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 657 (Actual)
Dates: Start 2010-07-06 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Diabetes | Time of examination
  Prevalence of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Hanson, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- Centro de Investigacion en Alimentacion y Desarollo (CIAD), Hermosillo, Mexico